CLINICAL TRIAL: NCT02451592
Title: SEIFEM 2015: Fungemia in Hematologic Malignancies
Brief Title: Fungemia in Hematologic Malignancies
Status: Completed | Type: Observational
Sponsor: Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne (Other)
Responsible Party: Principal Investigator, LIVIO PAGANO, MD, Hematology Professor, Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne
Other Study IDs: SEIFEM 2015
Record Dates: First submitted 2015-05-13; First posted 2015-05-22 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Acute Leukemia; Chronic Leukemia; Multiple Myeloma; Lymphoma
Keywords: Fungemia; Hematologic malignancies
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Fungemia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the risk factors for fungemia in a population of patients diagnosed with hematologic malignancies and eligible for chemotherapy.

DETAILED DESCRIPTION:
The coordinating center provides all participating centers with an epidemiologic form, in order to collect data in a comparable way. The requested informations include type of malignancy and its treatment, environmental expositions, laboratory work up, antifungal prophylaxis, clinical signs of infection, microbiological findings, antifungal therapy and outcome of infection at 30 days.

The planned sample size is about 300 patients to be recruited in 35 participating center over 5 years, in a retrospective-prospective fashion. Data check will be performed at the coordinating center. Missing data will be managed to minimize incomplete reports.

Statistical analysis will be performed by an independent reviewer, in order to assess risk factors predictive of fungal infection and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hematologic malignancies and eligible to chemotherapy

Exclusion Criteria:

* Patients not eligible to chemotherapy

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult and pediatric patients affected by hematologic malignancies and eligible to chemotherapy that develop fungemia
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Rate of fungemia outbreak during antifungal prophylaxis | Since 30 days average before fungemia onset

SECONDARY OUTCOMES:
Mortality from fungemia | After 30 days from fungemia onset

CONTACTS AND LOCATIONS:
Overall Officials: Livio Pagano, Professor, Principal Investigator — Catholic University of Sacred Heart, Rome Italy
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Pagano L, Caira M, Candoni A, Offidani M, Fianchi L, Martino B, Pastore D, Picardi M, Bonini A, Chierichini A, Fanci R, Caramatti C, Invernizzi R, Mattei D, Mitra ME, Melillo L, Aversa F, Van Lint MT, Falcucci P, Valentini CG, Girmenia C, Nosari A. The epidemiology of fungal infections in patients with hematologic malignancies: the SEIFEM-2004 study. Haematologica. 2006 Aug;91(8):1068-75. PMID 16885047
- [Background] Pagano L, Caira M, Nosari A, Van Lint MT, Candoni A, Offidani M, Aloisi T, Irrera G, Bonini A, Picardi M, Caramatti C, Invernizzi R, Mattei D, Melillo L, de Waure C, Reddiconto G, Fianchi L, Valentini CG, Girmenia C, Leone G, Aversa F. Fungal infections in recipients of hematopoietic stem cell transplants: results of the SEIFEM B-2004 study--Sorveglianza Epidemiologica Infezioni Fungine Nelle Emopatie Maligne. Clin Infect Dis. 2007 Nov 1;45(9):1161-70. doi: 10.1086/522189. Epub 2007 Sep 26. PMID 17918077
- [Background] Pagano L, Caira M, Candoni A, Aversa F, Castagnola C, Caramatti C, Cattaneo C, Delia M, De Paolis MR, Di Blasi R, Di Caprio L, Fanci R, Garzia M, Martino B, Melillo L, Mitra ME, Nadali G, Nosari A, Picardi M, Potenza L, Salutari P, Trecarichi EM, Tumbarello M, Verga L, Vianelli N, Busca A; SEIFEM Group. Evaluation of the practice of antifungal prophylaxis use in patients with newly diagnosed acute myeloid leukemia: results from the SEIFEM 2010-B registry. Clin Infect Dis. 2012 Dec;55(11):1515-21. doi: 10.1093/cid/cis773. Epub 2012 Sep 5. PMID 22955439
- [Background] Caira M, Candoni A, Verga L, Busca A, Delia M, Nosari A, Caramatti C, Castagnola C, Cattaneo C, Fanci R, Chierichini A, Melillo L, Mitra ME, Picardi M, Potenza L, Salutari P, Vianelli N, Facchini L, Cesarini M, De Paolis MR, Di Blasi R, Farina F, Venditti A, Ferrari A, Garzia M, Gasbarrino C, Invernizzi R, Lessi F, Manna A, Martino B, Nadali G, Offidani M, Paris L, Pavone V, Rossi G, Spadea A, Specchia G, Trecarichi EM, Vacca A, Cesaro S, Perriello V, Aversa F, Tumbarello M, Pagano L; SEIFEM Group (Sorveglianza Epidemiologica Infezioni Fungine in Emopatie Maligne). Pre-chemotherapy risk factors for invasive fungal diseases: prospective analysis of 1,192 patients with newly diagnosed acute myeloid leukemia (SEIFEM 2010-a multicenter study). Haematologica. 2015 Feb;100(2):284-92. doi: 10.3324/haematol.2014.113399. PMID 25638805
- [Background] Bassetti M, Merelli M, Righi E, Diaz-Martin A, Rosello EM, Luzzati R, Parra A, Trecarichi EM, Sanguinetti M, Posteraro B, Garnacho-Montero J, Sartor A, Rello J, Tumbarello M. Epidemiology, species distribution, antifungal susceptibility, and outcome of candidemia across five sites in Italy and Spain. J Clin Microbiol. 2013 Dec;51(12):4167-72. doi: 10.1128/JCM.01998-13. Epub 2013 Oct 9. PMID 24108614
- [Background] Pagano L, Fianchi L, Fanci R, Candoni A, Caira M, Posteraro B, Morselli M, Valentini CG, Farina G, Mitra ME, Offidani M, Sanguinetti M, Tosti ME, Nosari A, Leone G, Viale P. Caspofungin for the treatment of candidaemia in patients with haematological malignancies. Clin Microbiol Infect. 2010 Mar;16(3):298-301. doi: 10.1111/j.1469-0691.2009.02832.x. Epub 2009 Jun 22. PMID 19549221
- [Background] Pagano L, Antinori A, Ammassari A, Mele L, Nosari A, Melillo L, Martino B, Sanguinetti M, Equitani F, Nobile F, Carotenuto M, Morra E, Morace G, Leone G. Retrospective study of candidemia in patients with hematological malignancies. Clinical features, risk factors and outcome of 76 episodes. Eur J Haematol. 1999 Aug;63(2):77-85. doi: 10.1111/j.1600-0609.1999.tb01120.x. PMID 10480286
- [Background] Moore CB, Sayers N, Mosquera J, Slaven J, Denning DW. Antifungal drug resistance in Aspergillus. J Infect. 2000 Nov;41(3):203-20. doi: 10.1053/jinf.2000.0747. No abstract available. PMID 11120607
- [Background] Sanglard D, Odds FC. Resistance of Candida species to antifungal agents: molecular mechanisms and clinical consequences. Lancet Infect Dis. 2002 Feb;2(2):73-85. doi: 10.1016/s1473-3099(02)00181-0. PMID 11901654
- [Background] Nucci M, Marr KA, Vehreschild MJ, de Souza CA, Velasco E, Cappellano P, Carlesse F, Queiroz-Telles F, Sheppard DC, Kindo A, Cesaro S, Hamerschlak N, Solza C, Heinz WJ, Schaller M, Atalla A, Arikan-Akdagli S, Bertz H, Galvao Castro C Jr, Herbrecht R, Hoenigl M, Harter G, Hermansen NE, Josting A, Pagano L, Salles MJ, Mossad SB, Ogunc D, Pasqualotto AC, Araujo V, Troke PF, Lortholary O, Cornely OA, Anaissie E. Improvement in the outcome of invasive fusariosis in the last decade. Clin Microbiol Infect. 2014 Jun;20(6):580-5. doi: 10.1111/1469-0691.12409. Epub 2013 Nov 18. PMID 24118322
- [Background] Girmenia C, Pagano L, Martino B, D'Antonio D, Fanci R, Specchia G, Melillo L, Buelli M, Pizzarelli G, Venditti M, Martino P; GIMEMA Infection Program. Invasive infections caused by Trichosporon species and Geotrichum capitatum in patients with hematological malignancies: a retrospective multicenter study from Italy and review of the literature. J Clin Microbiol. 2005 Apr;43(4):1818-28. doi: 10.1128/JCM.43.4.1818-1828.2005. PMID 15815003